CLINICAL TRIAL: NCT03143413
Title: Ultrasonography Features of the Salivary Glands in Patient With Systemic Sclerosis: Comparison With Gougerot-Sjogren Syndrome and Sicca Asthenia Polyalgia Syndrome
Brief Title: Echo Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-323; 2016-A01256-45 (Other: 2016-A01256-45)
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Systemic Sclerosis; Gougerot Sjogren Syndrome; Sicca-Asthenia-Polyalgia Syndrome
Keywords: Salivary glands ultrasonography; Systemic sclerosis; Gougerot Sjogren syndrome; Sicca syndrome
MeSH Terms: conditions — Scleroderma, Systemic; Sjogren's Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Systemic sclerosis: Systemic sclerosis is an autoimmune connective tissue disease with undefined etiology and characterized by progressive fibrosis of the skin and major organs. Dry eyes and / or buccal syndrome is commonly reported in patients with systemic sclerosis.
  Interventions: Other: Ultrasonography
- Gougerot-Sjogren syndrome: Goujerot-Sjogren syndrome is a chronic autoimmune disorder that is characterized by dryness of the eyes (xerophthalmia) and / or mouth (xerostomia).
  Interventions: Other: Ultrasonography
- Sicca-Asthenia-Polyalgia syndrome: It may be primary or secondary to another connective tissue disease (such as lupus, rheumatoid arthritis or other).
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — Patient will be enrolled in the rheumatology department of University hospital of Clermont-Ferrand (France).
  Salivary glands ultrasonography will be performed on all patients enrolled by the same expert and blinded to the diagnosis of the patient. Echostructure of the two salivary glands will be graded 0 to 4 and the size calculated.

SUMMARY:
Systemic sclerosis is an autoimmune connective tissue disease with undefined etiology and characterized by progressive fibrosis of the skin and major organs. Dry eyes and / or buccal syndrome is commonly reported in patients with systemic sclerosis. Goujerot-Sjogren syndrome is a chronic autoimmune disorder that is characterized by dryness of the eyes (xerophthalmia) and / or mouth (xerostomia). It may be primary or secondary to another connective tissue disease (such as lupus, rheumatoid arthritis or other). Several criteria have been validated to classify the SS but require a labial salivary gland biopsy, invasive act which complications can sometimes be reported (hematoma, lip sensory defect).

Several scores based on the evaluation of the ultrasound homogeneity of the salivary glands were developed but no studies have evaluated ultrasound abnormalities of salivary glands in patients with systemic sclerosis.

DETAILED DESCRIPTION:
Descriptive explorative study of three population showing sicca symptoms (Systemic sclerosis, Gougerot-Sjogren syndrome, Sicca-Asthenia-Polyalgia syndrome).

Patient will be enrolled in the rheumatology department of University hospital of Clermont-Ferrand (France).

Salivary glands ultrasonography will be performed on all patients enrolled by the same expert and blinded to the diagnosis of the patient. Echostructure of the two salivary glands will be graded 0 to 4 and the size calculated.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis diagnosis established by a rheumatologist and met ACR 2012 criteria
* Or primary Gougerot-Sjogren patient who met American-European Consensus Group (AECG) classification criteria.
* Or patient presenting a sicca syndrome but not met Gougerot-Sjogren criteria

Exclusion Criteria:

* History of radiotherapy on face and neck
* Infection such as VIH or Hepatitis C
* Sarcoidosis
* Amylosis
* Wearing contact lenses
* Hyper IgG4 syndrome

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 20 systemic sclerosis, 40 Gougerot-Sjogren syndrome, 40 Sicca-Asthenia-Polyalgia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Jousse-Joulin ultrasonography score | the day of inclusion
  Echostructure of the two salivary glands will be graded 0 to 4 and the size calculated.

SECONDARY OUTCOMES:
Ultrasonography score equal or higher than 2 on at least one salivary gland | the day of inclusion
Ultrasonography score equal or higher than 3 on at least one salivary gland | the day of inclusion
Global ultrasonography score higher than 6/16 | the day of inclusion
Salivary glands area | the day of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France